CLINICAL TRIAL: NCT00670995
Title: Tobacco World: Interactive Tobacco Education for Teens
Brief Title: Tobacco Zero: Interactive Tobacco Education for Teens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deschutes Research, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103623B
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco use among middle and junior high school students remains a concern among health educators.; The use of tobacco prevention programs and their integration into school-based curricula has been lacking due to a number of factors.
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Interactive Tobacco Education — Increase perceived behavioral control (self-efficacy) Decrease willingness to use tobacco Decrease intentions to use tobacco

SUMMARY:
There have been a number of tobacco prevention programs developed and tested in the past few years, and some of the comprehensive programs have been promoted by the Office on Smoking and Health at the Centers for Disease Control (CDC). However, the use of these programs and integration into school-based curriculum has been lacking due to a number of factors. We are proposing to develop an interactive computer-based program for tobacco prevention aimed at middle school students. The CD-ROM is designed to be an adjunct to the existing health education curriculum provided for 6th through 8th grade students.

DETAILED DESCRIPTION:
The CD-ROM is based upon our Phase I prototype program entitled Tobacco World in which students are presented with a video arcade interface that offers them random access to several game-like activities in which they learn about tobacco and the negative health effects associated with tobacco use. We will expand the menu of options to include more complex activities and entertaining games.

The Phase II program will deliver engaging media to educate students about the risks of tobacco and peer and industry influences on their decisions regarding tobacco. Games and activities will be designed to act on mechanisms shown to be effective in decreasing intentions to use tobacco through changing attitudes, social images, beliefs about short and long term physical consequences, perceptions of peers' social images, subjective norms, and perceived behavioral control. We will test individual components of the program with middle school students for effectiveness in changing mediating variables related to initiation and use of tobacco.

The final program will be evaluated in a randomized trial where middle schools in Oregon and New York will be assigned to either an established tobacco prevention curriculum, or to the usual tobacco curriculum plus the Tobacco World program. Students will be assessed at pre-, post- and 6-month follow-up to evaluate the impact of program use on intentions, and actual tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Middle school students in 6th or 7th or 8th grade in Oregon and New York City whose parents have consented to have their child participate;
* Middle school health education teachers in Oregon and New York City

Exclusion Criteria:

* Students unable to understand English.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1864 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Increase perceived behavioral control (self-efficacy) | pre and post

SECONDARY OUTCOMES:
Decrease willingness to use tobacco | pre and post
Decrease intentions to use tobacco | pre and post

CONTACTS AND LOCATIONS:
Overall Officials: Herbert H Severson, PhD, Principal Investigator — Deschutes Research, Inc.
Locations (1):
- Deschutes Research Inc, Eugene, Oregon, United States